CLINICAL TRIAL: NCT05872113
Title: Product A (Test Product), Product B (Control Product) Evaluation of Human Efficacy for Skin Moisturization and Wrinkle Improvement
Brief Title: Evaluation of Human Efficacy for Skin Moisturization and Wrinkle Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ji Hye Yoon (Other)
Collaborators: COSMAX (Unknown); Global medical research center (Unknown)
Responsible Party: Sponsor-Investigator, Ji Hye Yoon, Principal Investigator, Sungkyunkwan University
Organization: Sungkyunkwan University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: GIRB-21929-NY
Record Dates: First submitted 2023-03-28; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Dry Skin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): The subjects who were on a placebo were put on the cream two times per day for 4 weeks. The questionnaire for testing the effects progressed when before using the cream, after 2 weeks, and after 4 weeks.
  Interventions: Combination Product: Placebo cream
- Experiment (Experimental): The subjects who were on experimental were put on the cream two times per day for 4 weeks. The questionnaire for testing the effects progressed when before using the cream, after 2 weeks, and after 4 weeks.
  Interventions: Combination Product: Hs-hWE cream

INTERVENTIONS:
Combination Product: Hs-hWE cream — The cream was applied to the faces of subjects, the left facial area was put on the 0.5% Hs-WE cream.
  Arms: Experiment
Combination Product: Placebo cream — The cream was applied to the faces of subjects, the right facial area was put on the placebo cream.
  Arms: Placebo

SUMMARY:
All subjects used the placebo sample on the left side of their face and the investigational sample on the right side of their face, respectively. The moisturizing levels were detected before use (0 week), after 2 weeks and after 4 weeks. The wrinkles of subjects were also measured on the same date interval as the skin moisture level test.

DETAILED DESCRIPTION:
Twenty-two subjects were initially enrolled in the clinical trial. One subject was excluded by non-compliance with the plan of trials. All subjects used the placebo sample on the left side of their face and the investigational sample on the right side of their face, respectively. The moisturizing levels were detected before use (0 week), after 2 weeks and after 4 weeks. The crow's feet of subjects were also measured on the same date interval as the skin moisture level test.

ELIGIBILITY:
Inclusion Criteria:

* Females with dried skin, aged 30-59 years (average=49.2 yrs).
* The subject has eye wrinkles (crow's feet).
* A person who has voluntarily signed consent after fully explaining the test purpose and content.
* Those who can follow up during the test period.
* A healthy person without acute or chronic physical disease including skin disease.

Exclusion Criteria:

* Pregnant or lactating women and women of childbearing age who do not agree to the contraceptive method prescribed by the protocol.
* A person with a lesion at the test site or suffering from an infectious skin disease.
* People with allergies or hypersensitivity, or irritation to cosmetics, pharmaceuticals, or daily exposure to light.
* Those who have received systemic steroids or phototherapy within 1 month of participating in the trial, or who have received skin treatment (scaling/botox/filler/laser/tattoo) within 3 months of participating in the trial.
* Those who have used drugs with similar functions at the research site within 3 months before the start of the study, or have a mental illness, or mental retardation disorder.
* Other than the above, a person who will make it difficult to conduct a human test based on the judgment of the responsible researcher or the person in charge of the study.

Ages: 30 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Evaluation of Human Efficacy for Skin Moisturization Improvement through visual assessment | up to 4 weeks
  The skin moisture level of subjects were also measured on the 0, 2, 4 weeks. skin moisturizing level was conducted using a Corneometer CM825 (Courage and Khazaka, Köln, Germany). The measurement of skin moisturization used capacitance, and the difference in dielectric constant between water and the measuring material was expressed as a measured value.
Evaluation of Human Efficacy for skin Wrinkle Improvement through visual assessment | up to 4 weeks
  The skin wrinkles of subjects were measured on the 0, 2, and 4 weeks. Skin wrinkles were approximated by visual assessment using an Antera 3D CS (Miravex, Ireland). The depth (Depth, mm) image of the Wrinkle-small analysis mode was used as evaluation data for skin wrinkle measurement. The measuring device was a device that can measure the condition of the skin's epidermis and dermis using a light emitting diode (LED light source), extract data from three-dimensional shape images, quantify skin conditions, and monitor skin changes over time to measure skin wrinkles.

CONTACTS AND LOCATIONS:
Locations (1):
- Sungkyunkwan university, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: Yes